CLINICAL TRIAL: NCT01733537
Title: Improving Motorcycle Taxi Driver Visibility in Tanzania-A Cluster Randomized Controlled Trial
Brief Title: Improving Motorcycle Taxi Driver Visibility in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00034415; 1R25TW009337-01 (NIH)
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Accidents, Traffic
Keywords: traffic accidents, motorcycle, injury, conspicuity
MeSH Terms: conditions — Wounds and Injuries | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vest and Education (Experimental): Motorcycle Taxi Drivers provided with a reflective, fluorescent vest and basic education about recommended measures to increase their visibility
  Interventions: Other: Free reflective, fluorescent vest; Behavioral: Education
- Education Alone (Other): Motorcycle Taxi Drivers provided with basic education about recommended measures to increase their visibility
  Interventions: Behavioral: Education

INTERVENTIONS:
Other: Free reflective, fluorescent vest — Motorcycle taxi drivers in the intervention arm will receive a free reflective, fluorescent vest
  Arms: Vest and Education
Behavioral: Education — Both arms will receive brief, basic education about recommended measures to increase their visibility

SUMMARY:
The purpose of this study is to determine whether providing motorcycle taxi drivers with a free reflective fluorescent vest will result in increased use of reflective or fluorescent clothing compared to education about wearing reflective or fluorescent clothing alone.

DETAILED DESCRIPTION:
Road traffic injuries are the 4th leading cause of death among individuals in the economically productive age group (age 15 to 59) in low and middle income countries. The Africa region currently has some of the world's highest traffic injury rates, with vulnerable road users, including motorcycle riders, bearing a disproportionate share of the injury burden.

Motorcycles are a rapidly growing form of transport in Africa, both for personal and commercial transportation. Conspicuity measures-factors that increase a motorcycle rider's visibility-for the prevention of motorcycle crash have been previously studied and found to be associated with a decreased risk of crash.

Motorcycle taxi drivers are a particularly high risk population for motorcycle crash as they operate a motorcycle for several hours a day. Reflective, fluorescent safety vests are a common article worn by motorcycle drivers in some locations; however, penetration of such clothing in Moshi is currently low. This study aims to increase use of reflective vests among commercial motorcycle drivers. We will test whether provision of a free reflective, fluorescent vest increases use of reflective, fluorescent clothing compared to education about wearing reflective, fluorescent clothing alone.

ELIGIBILITY:
Inclusion Criteria:

* motorcycle riders who identify themselves as motorcycle taxi drivers
* individuals must work at least 2 days a week as a motorcycle taxi driver
* have a telephone number for ride solicitation
* have a license plate that is able to be recorded
* are at least 18 years old
* are willing to have us contact them in the future for repeat surveys

Exclusion Criteria:

* motorcycle riders who do not meet the above criteria
* motorcycle riders who do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Use of reflective or fluorescent clothing | 3-5 months
  The use of reflective or fluorescent clothing will be compared between the intervention and control groups over the observation period

SECONDARY OUTCOMES:
Wearing White Helmet | 3-5 months
  The use of white helmets will be compared between the intervention and control groups over the observation period
Daytime Running Headlights | 3-5 months
  The use of daytime running headlights will be compared between the intervention and control groups over the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Nathan M Thielman, MD, MPH, Principal Investigator — Duke University; Steven A Sumner, MD, Study Director — Duke University
Locations (1):
- Kilimanjaro Region, Tanzania, Kilimanjaro Region, Kilimanjaro, Tanzania